CLINICAL TRIAL: NCT01891617
Title: The Exercise Effects on Appetite and Gut Peptides While on High-fat Diet
Brief Title: Exercise Effects on Insulin, Gut Peptides, and Appetite
Acronym: XFG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Dr. Katarina Borer, Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R15DK082800-XFG; R15DK082800 (NIH)
Record Dates: First submitted 2013-06-26; First posted 2013-07-03 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Endocrine and Metabolic Responses to Exercise and Diets
Keywords: exercise; high carbohydrate and high fat diets; insulin; gut peptides; appetite; metabolism; glucose
MeSH Terms: conditions — Motor Activity; Insulin Resistance | interventions — Exercise; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exercise-high-fat diet (Experimental): Two bouts of exercise followed by a high-fat meal
  Interventions: Other: Exercise and diets
- Exercise-high-carbohydrate diet (Experimental): Two bouts of exercise followed by a high-carbohydrate meal
  Interventions: Other: Exercise and diets
- Sedentary-high-fat diet (Experimental): Sedentary trial with two high-fat meals
  Interventions: Other: Exercise and diets
- Sedentary-high-carbohydrate diet (Experimental): Sedentary trial with two high-carbohydrate meals
  Interventions: Other: Exercise and diets

INTERVENTIONS:
Other: Exercise and diets — Exercise and high-fat diet Exercise and high-carbohydrate diet Sedentary and high-fat diet Sedentary and high-carbohydrate diet

SUMMARY:
Determine whether the mid-day suppression of hunger and amplified increase in the release of glucose-dependent insulinotropic peptide (GIP) and glucagon-like peptide 1 (GLP-1) following morning exercise is due to increased fat content of the diet per se or a combination of high fat diet after morning exercise. The action of gut peptides, particularly GLP-1, on gastric emptying is likely to be important in mediating its effects on postprandial appetite and glycemia (Nauck et al. 1997). Our hypothesis is that exercise amplifies gut peptide secretion when diet is enriched with fat, and that this stimulus suppresses the hunger sensation.

DETAILED DESCRIPTION:
Specific aim: Determine whether a change in macronutrient composition from 60% carbohydrate and 25% fat to 30% carbohydrate and 45% fat is responsible by itself for suppression of hunger and increased secretory response of glucose-dependent insulinotropic hormone (GIP) and glucagon-like peptide-1 (GLP-1), or whether these changes depend on preceding exercise. We will measure (a) concentrations of plasma GIP and GLP-1 by chemiluminescent multiplex assay, (b) concentrations of plasma ancetaminophen to assess the gastric emptying rate, (c) concentrations of plasma insulin, and glucagon by radioimmunoassay, and glucose, ketone bodies, and free fatty acids with appropriate spectrophotometric methods, (d) hourly appetite responses with visual analog scale under two conditions: sedentary (SED) and exercise (EX).

Hypothesis: Hunger suppression and secretion of GIP and GLP-1 after the morning meal will be greater with slower gastric emptying rate when a meal consisting of 45% fat and 30% carbohydrate follows three hours after a 2-hour bout of moderate-intensity exercise than in the absence of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal status
* Age 50 to 65 years
* BMI between 20 and 30 kg/m2.
* Good health status (normotensive, fasting glucose < 100 mg/dl, , hematocrit > 32%, hemoglobin >12 mg/dl)
* Absence of restricted food intake
* Absence of endocrine and metabolic disorders requiring medication other than hormonally corrected hypothyroidism
* Absence of musculoskeletal disabilities that would prevent walking

Exclusion Criteria:

* Presence of endocrine and metabolic disease requiring medication, other than hormonally corrected hypothyroidism
* Presence of musculoskeletal disabilities that would prevent walking
* Smoking
* Active dieting
* Absence of listed inclusion criteria
* Unwillingness to follow study protocol.

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-11; Primary Completion 2012-07 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Plasma insulin concentration | 36 hours
  Change in plasma insulin to two bouts of exercise followed by a high-carbohydrate or a high fat diet
Plasma glucagon concentration | 36 hours
  Changes in plasma glucagon concentration to two bouts of exercise followed by either a high-carbohydrate or a high-fat meal
Plasma concentration of glucose-dependent insulinotropic peptide (GIP) | 36 hours
  Changes in plasma concentration of glucose-dependent insulinotropic peptide (GIP)to two bouts of exercise followed by either a high-carbohydrate or a high-fat meal
Plasma concentration of free fatty acids | 36 hours
  Changes in plasma concentration of free fatty acidsto two bouts of exercise followed by either a high-carbohydrate or a high-fat meal
Plasma concentration of beta-hydroxybutyrate | 36 hours
  Changes in plasma concentration of beta-hydroxybutyrate to two bouts of exercise followed by either a high-carbohydrate or a high-fat meal
Plasma glucose concentration | 36 hours
  Changes in plasma glucose concentration to two bouts of exercise followed by either a high-carbohydrate or a high-fat meal
daytime hourly appetite ratings | 36 hours
  Changes in daytime hourly appetite ratings to two bouts of exercise followed by either a high-carbohydrate or a high-fat meal

SECONDARY OUTCOMES:
Plasma concentrations of glucagon-like peptide-1 (GLP-1) | 36 hours
  Changes in plasma concentrations of glucagon-like peptide-1 (GLP-1)to two bouts of exercise followed by either a high-carbohydrate or a high-fat meal
Plasma concentrations of peptide tyrosine tyrosine (PYY) | 36 hours
  Changes in plasma concentrations of peptide tyrosine tyrosine (PYY) to two bouts of exercise followed by either a high-carbohydrate or a high-fat meal

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Borer, PhD, Principal Investigator — University of Michigan
Locations (1):
- Michigan Clinical Research Unit, Ann Arbor, Michigan, United States